CLINICAL TRIAL: NCT06723626
Title: Clinical Study of the Effect of Intravenous Hydrocortisone Combined With Vitamin C and Vitamin B1 Infusion on Prognosis and Sublingual Microcirculation in Elderly Patients With Sepsis or Septic Shock.
Brief Title: Effects of Intravenous Metabolic Recovery Agent in Elderly Septic Patients on Prognosis and Microcirculation.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Southeast University, China (Other)
Responsible Party: Principal Investigator, Jingyuan,Xu, Clinical Professor, Southeast University, China
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2023ZDSYLL355-P01
Record Dates: First submitted 2024-05-21; First posted 2024-12-09 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Septic Shock
Keywords: hydrocortisone; vitamin C; vitamin B1; sepsis; septic shock; mortality; microcirculation
MeSH Terms: conditions — Shock, Septic; Sepsis | interventions — Hydrocortisone; Ascorbic Acid; Thiamine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- metabolic resuscitation agents (Experimental): Patients in the intervention group received IV hydrocortisone (200mg every 24 hours), vitamin C (1.5g every 6 hours), and thiamine (200 mg every 12 hours).
  Interventions: Drug: Metabolic resuscitation agent
- hydrocortisone (Placebo Comparator): Patients in the control group received IV hydrocortisone (200mg every 24 hours).
  Interventions: Drug: Hydrocortisone

INTERVENTIONS:
Drug: Metabolic resuscitation agent — Intervention group will receive intravenous hydrocortisone (200mg every 24 hours), vitamin C (1.5g every 6 hours), and thiamine (200 mg every 12 hours).
  Other Names: Hydrocortisone, vitamin C and vitamin B1
  Arms: metabolic resuscitation agents
Drug: Hydrocortisone — Placebo group will receive intravenous hydrocortisone 200mg every 24 hours.
  Arms: hydrocortisone

SUMMARY:
This study intends to observe the effect of intravenous hydrocortisone combined with vitamin C and vitamin B1 infusion on the prognosis and sublingual microcirculation in patients with sepsis or septic shock through a prospective randomized controlled study method.

DETAILED DESCRIPTION:
Shock is a common pathophysiological state in critical care medicine and occupies an important position. In recent years, some studies have had uesd metabolic resuscitation agent -- namely hydrocortisone + vitamin C + vitamin B1 cocktail therapy in the treatment of sepsis patients, studies found that this method may reduce the lactate level, improve renal failure and circulatory failure, and then improve the prognosis of such patients. There are also study groups that do not significantly prolong the survival of septic shock, suggesting that we need to screen out the use of metabolic resuscitation agents. Given the important role of vitamins in shock, uncontrolled inflammatory response, capillary leakage, and microcirculation dysfunction, whether the improved prognosis may be related to the patients' own vitamin levels. Vitamin deficiency is often present in the elderly.

This study aims to observe the effect of precision treatment of metabolic resuscitation agent on mortality and sublingual microcirculation in the follow-up prognosis of elderly septic patients on the basis of monitoring vitamin B1 and C levels in elderly septic patients.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥60 and ≤85 years old;
* Diagnosis of sepsis or septic shock;
* Clinical judgment for hydrocortisone treatment;
* Signing Informed Consent.

Exclusion Criteria:

* patients in palliative care;
* uncontrolled malignancy with multiple metastases;
* ineffective surgical intervention for the infectious agent;
* estimated death within 24 hours;
* glucocorticoids used in the last 7 days;
* allergy to hydrocortisone, vitamin c or vitamin B1;
* inability to measure sublingual microcirculation.

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
28-d Mortality | 28 days after treatment
  patients with sepsis who died after treatment from any cause within 28 days

SECONDARY OUTCOMES:
Perfused vessel density (PVD) | 48 hours after treatment
  Determinant of capillary diffusive capacity
proportion of perfusion vessels | 48 hours after treatment
  sublingual microcirculation parameter
Lactate clearance, 48h, % | 48 hours after treatment
  Tissue perfusion parameter

CONTACTS AND LOCATIONS:
Overall Officials: Jingyuan Xu, M.D., Principal Investigator — Zhongda Hospital
Locations (1):
- Zhongda Hospital Southeast University, Nanjing, Jiangsu, China